Development of methods and algorithms for diet design based on gut microbiota analysis

# Study protocol

Number of clinical trial: 1631

**Project number: NSP67** 

Approved by Ethical Committe of National Institute for Health Development 25.10.2016

"Development of methods and algorithms for diet design based on gut microbiota analysis"

#### Study protocol

#### **General plan**

Time Activity

Day 1, 2 ... 31 Food diary (at least 3 days before fecal sampling)

Day 1 Questionnaire about health conditions

Day 4 and 32 Faecal sampling, Bristol and bowel habit estimation

Sending sample to the lab

Weight measurement

### **Activity plan**

- Start keeping a food diary, 3 days before the first faecal sample is collected. Keep a diary (on paper, in a word processor, or in a web-based nutrition program) of everything you drove and drank during the day (including any breaks).
  - 2. Fill in the questionnaire (on paper, in a word processing program or online).
  - 3. On day 4 take a sample of the faeces using both the spoon method and the cotton swab method (instructions below).
- 4. Send samples just after the sampling to the lab using the storage box placed in the sending box labelled with address.
  - 5. Start keeping the diet plan according to the instructions provided by the nutritionist.
- 6. On day 32 take a sample of the faeces using both the spoon method and the cotton swab method (instructions below).
- 7. Send samples just after the sampling to the lab using the storage box placed in the sending box labelled with address.

#### Instruction for faecal sampling

- 1. Use FecesCatcher for faecal sampling.
- 2. Stick the FecesCatcher paper collector on the back of the toilet seat with self-adhesive edges (NB! Do not touch the waterline, see illustrated instruction on the separate sheet provided).
  - 3. Avoid getting urine (and water) in the FecesCatcher, as this can cause the paper to break.
    - 4. Collect the stool on paper so that it does not mix with urine.
  - 5. Evaluate the consistency of the faeces using the Bristol scale and the color of the faeces.

    Mark this on the attached sheet.
    - 6. Take a sample of the faeces using both
    - a. the spoon method (follow the detailed instructions provided on the separate sheet)



b. the cotton swab method (follow the detailed instructions provided on the separate



## sheet)

- 7. After sampling, release the FecesCatcher from the toilet seat, press the edges together, and allow them to fall into the pot and flush down
  - 8. Video instruction: https://www.youtube.com/watch?v=hsAyURaBKv0